CLINICAL TRIAL: NCT03519100
Title: Rhinoplasty and Quality of Life: Prospective Multicenter Study Before and After Surgery
Brief Title: Rhinoplasty and Quality of Life
Acronym: FACE-Q
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/40
Record Dates: First submitted 2018-04-05; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Rhinoplasty; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of life evaluation — quality of life evaluation post surgery

SUMMARY:
Quality of life and satisfaction in aesthetic surgery is still under-evaluated. It is a prospective and multicenter study with a 4 months follow-up of patients under rhinoplasty or rhinoseptoplasty procedure. They will answer to the FACE-Q and NOSE questionnaires before surgery, one week later and 4 months after the procedure. The aim of the study is to show a significant augmentation of the quality of life scores. At this occasion, the FACE-Q questionnaire has been translated and validated in French

DETAILED DESCRIPTION:
The main objective of this study is to show the efficiency of the rhinoplasty or rhinoseptoplasty procedure on the quality of life in a French population. There are many Patients reported outcomes questionnaire in aesthetic surgery but none of them is perfect. The FACE-Q rhinoplasty modules questionnaires is a recent test which has been validated in English but not in French. It is able to evaluate different areas of the quality of life and patient satisfaction. After French validation of the FACE-Q, this study will compare patient satisfaction before and after rhinoplasty or rhinoseptoplasty procedure. There is a lack of studies in the French population about rhinoseptoplasty surgery and quality of life or satisfaction. The goal is to show the interest of a surgery procedure on the feeling of the patients, concerning very different domains of appearance. This could help us to define the preoperative patients who are able to be really improved by this surgery

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old,
* patient engaged for surgery procedure of rhinoplasty or rhinoseptoplasty

Exclusion Criteria:

* patient with nose surgery medical history,
* mental or physical incapacity to answer the questionnaires
* antecedent of cervico facial cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will involved during surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change between the FACE-Q score | at the inclusion, one week later and 4 months after surgery
  Change between the FACE-Q score at the inclusion, one week later and 4 months after surgery. The minimal clinical importance difference has to be determinate thanks to the validation process of the FACE-Q in French

SECONDARY OUTCOMES:
Difference between the NOSE score | at the inclusion and 4 months post surgery
  Difference between the NOSE score at the inclusion and 4 months after surgery
Difference between anthropometrics measures | before and immediate post surgery
  Difference between anthropometrics measures of the nose before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: de GABORY Ludovic, Study Director — University Hospital, Bordeaux
Locations (1):
- UH Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No